## **Cover Page**

Official Title of the Study: Validation of Point Partial User Needs With Partial Finger

Amputees

Document Date: October 22, 2019

NCT Number: NCT05012657

## **Statistical Analysis Plan**

This is not a statistically powered study. This is a device feasibility test with pass/fail results for objective tasks. The validation methods described in Table 1 will be implemented to confirm the user needs of the *Point Partial*. A simple pass/fail result will be recorded for each user need for each subject. No formal outcome measures nor data analysis will be performed during this sub-aim (a statistically powered study is presented in Aim #2.2). Here, we are focused on confirming that the product suits our user needs in its first use by human subjects. An overall passing rate above 80% across all user needs and subjects will be considered a success.

Table 2. User Needs and Validation Methods for Point Partial

| User Need | | Validation Method | |
|---|---|---|---|
| ID# | Description | ID# | Description |
| UN-1 | Point Partial shall be comfortable for a full day's use | VAL-1 | User wears <i>Point Partial(s)</i> for a full day |
| UN-2 | Point Partial shall allow the user to flex and extend finger without their contralateral hand | VAL-2 | User flexes and extends the <i>Point</i> Partial(s) without using contralateral hand |
| UN-3 | Point Partial shall be robust enough to operate in challenging environments | VAL-3.1 | User lifts a 25 lb. bag with <i>Point</i> Partial(s) |
| | | VAL-3.2 | User grips a hammer with <i>Point</i> Partial(s) and drives a nail into a piece of wood |
| UN-4 | Point Partial shall be releasable while performing active grasps | VAL-4 | User releases <i>Point Partial(s)</i> while performing an active grasp by pressing the dorsal button |
| UN-5 | Point Partial shall have a durable ratcheting mechanism | VAL-5 | User positions <i>Point Partial(s)</i> into each of the locking positions |
| UN-6 | Point Partial shall have a reliable auto spring-back mechanism | VAL-6 | User activates spring-back mechanism by using (1) contralateral hand, (2) tabletop, and (3) side or thigh |
| UN-7 | Point Partial shall have high friction | VAL-7 | User grips a 5 lb. cylindrical smooth object using <i>Point Partial(s)</i> for 10 seconds |
| UN-8 | Point Partial shall have a pronounced fingernail | VAL-8 | User picks up 1 coin from a smooth tabletop |
| UN-9 | Point Partial shall be robustly attached to mounting system | VAL-9 | User performs VAL-1 through VAL-8 |